CLINICAL TRIAL: NCT03466957
Title: Development and Assessment of Individual 3D Printed Applicators in MRI Guided Gynecological Brachytherapy
Brief Title: Individual Approach in Gynecological Cancer Brachytherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERID-KESOPKR/63
Record Dates: First submitted 2018-03-01; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Cancer
Keywords: image guided brachytherapy; 3D print; gynecological cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D printed applicator (Experimental): individually designed applicator for BT
  Interventions: Other: 3D printed applicator

INTERVENTIONS:
Other: 3D printed applicator — add-on cap for oblique needles, 3D printed Vienna-like applicator, individual vaginal cylinder for intracavitary/interstitial application
  Other Names: individual applicator

SUMMARY:
MRI guided adaptive brachytherapy (BT) represents the gold standard in the treatment of gynecological cancers. Commercially available standard MRI compatible applicators for BT of gynecological cancers don't always allow for optimal target volume coverage. Three-dimensional (3D) printed technology enables versatile possibilities of improvement of standard applicators and development of novel applicators with better coverage of the target volume. The purpose of this study is to implement and assess 3D printing technology as an instrument for designing and manufacturing applicators for individualized BT of gynecological cancers.

DETAILED DESCRIPTION:
Patients with locoregionally gynecological cancers will be included in this single-institution, non-randomized, one-arm study. All patients will receive 45-50 Gy external beam radiotherapy (EBRT) with intensity-modulated radiotherapy/volumetric-modulated arc therapy (IMRT/VMAT) technique, 1.8-2 Gy/fraction +/- concurrent cisplatin based chemotherapy. First BT with commercially available standard applicators (tandem with ring +/- parallel needles or vaginal cylinder) will be carried out. MRI with applicator in situ will be performed, high-risk clinical target volume (CTV-HR) and organs at risk (OAR) will be delineated and treatment planning will be conducted. In the case of large gynecological cancer and suboptimal target coverage at BT (V100 ≤ 90%, D98 ≤ 80%, D90 ≤ 100%, D100 ≤ 60%) a preplan will be performed as the basis for the 3D applicator modelling. The next BT application will be performed with an individually designed 3D printed applicator. Dose-volume characteristics of the following treatment plans will be compared: the preplan, the plan with standard and the plan with individual 3D printed applicator.

The primary objective of the study is to determine the improvement of dose-volume parameters with the use of 3D printed individual applicators in advanced gynecological cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with locally advanced gynecological cancer (cervical, uterine, vaginal, vulvar cancer) eligible for treatment with brachytherapy
* squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma, histologically proven
* patients fit for regional or general anesthesia
* signed written informed consent

Exclusion Criteria:

* regional or general anesthesia contraindications
* contraindications for MRI

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
target volume CTV-HR | at two hours after the end of brachytherapy procedure
  V100 (%), D90 (%), D98 (%), D100 (%)

SECONDARY OUTCOMES:
organs at risk | at two hours after the end of brachytherapy procedure
  D2cc (Gy), D0.1cc (Gy), Dmax (Gy)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Barbara Zobec Logar, MD, Principal Investigator — Brachytherapy Department, Institute of Oncology Ljubljana, Slovenia
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia